CLINICAL TRIAL: NCT05192096
Title: Capacity Building and Service Enhancement of Integrated Home Care Services During COVID-19
Brief Title: Capacity Building and Service Enhancement in Integrated Home Care Services
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Aberdeen Kai-fong Welfare Association (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant professor, The University of Hong Kong
Other Study IDs: UW21-781
Record Dates: First submitted 2021-12-29; First posted 2022-01-14 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: COVID-19, risk management, service enhancement, capability building
MeSH Terms: conditions — Behavior; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention group: It includes two 1-hour health-related information sessions.
  Interventions: Behavioral: Train-the-trainer workshop

INTERVENTIONS:
Behavioral: Train-the-trainer workshop — To deliver health-related information to trainees, which facilitate improving their knowledge, confidence, and ability to share and discuss health-related information with others, including service users, families and friends.

SUMMARY:
As people live longer lives, the ageing population causes an unprecedented rise in healthcare and social services demand. Limited studies were to evaluate the effectiveness of risk management measures of home care service and the needs of service workers, which raised concerns about the needs of staff working in home care settings and how service organizations continuously dealt with those challenges in this ongoing pandemic.

This study includes two parts: Part 1, Needs assessment, a survey to collect feedback from staff and understand their needs.; Part 2, Train-the-trainer workshops for staff and volunteers as lay health promoters to build workforce capacity and enhance trainees' competence and performance in delivering brief health-related information to their service users during COVID-19. It includes quantitative questionnaire assessment and qualitative focus group interview.

DETAILED DESCRIPTION:
With modern medicine and technological advancements, the global life expectancy has increased over the last century. As people live longer lives, the ageing population causes an unprecedented rise in demand for healthcare and social services. Integrated Home Care Services (IHCS) provides care and community support services to elderly persons and people with disabilities according to their individual and social needs, to enable them to continue living in the community. This approach helps maintain a sense of attachment and feelings of security and familiarity in relation to both homes and communities and reduces the overload of nursing homes.

The Aberdeen Kai-fong Welfare Association Social Service (AKA) is one of the 61 non-government organisations (NGO) under the IHCS. AKA provides a wide range of services which include home care, nursing and rehabilitation services for elders, people with disabilities and families in need (service users) in the Southern District of Hong Kong.

The pandemic of COVID-19 has brought significant challenges globally and locally. With the safety and distancing measures from the government, the scope of Integrated Home Care Services was restricted to essential services during the early stage of the pandemic. Apart from the suspension of services, other major challenges of home care service providers faced were an insufficient supply of personal protective equipment, an insufficient workforce, inadequate training. These problems have all led to infection control concerns for home care institutions and their staff. To combat the spread of the virus and maintain the continuity of services, IHCS providers applied a series of risk management measures throughout the pandemic.

The train-the-trainer (TTT) model is gaining increasing attention as an effective strategy to build a community workforce for health promotion and disease prevention. Training for participants from the same community they serve as lay health promoters (volunteers), can help build knowledge at the local level. Lay health promoters with training and supervision were shown to have significant impacts on community-based interventions. The training of lay health promoters and reliance on community resources simultaneously reduce the demand on time, resources and manpower from financially strapped and understaffed professional social health services in the community.

Limited studies were to evaluate the effectiveness of risk management measures of home care service and the needs of service workers, which raised concerns about the needs of staff working in home care settings and how service organizations continuously dealt with those challenges in this ongoing pandemic. Besides, the lack of training programs was systematically evaluated.

This proposed study includes two parts: Part 1, Need assessment, a survey to collect feedback from staff and understand their needs.; Part 2, Train-the-trainer workshops for staff and volunteers as lay health promoters to build workforce capacity and enhance trainees' competence and performance in delivering brief health-related information to their service users during COVID-19. Questionnaire assessments will be conducted at baseline, immediately after each session, one- and three-month follow up. Focus-group interviews will be conducted at the end of the study (completion of all train-the-trainer workshops and assessments).

ELIGIBILITY:
Part 1: Needs assessment

Inclusion criteria

• Staff of Aberdeen Kai-fong Welfare Association under the division of Integrated Home Care Services

Exclusion criteria

* Subjects refuse to answer this questionnaire
* Subjects who are unable to read and understand Chinese

Part 2: Train-the-trainer workshops

Inclusion criteria

• Staff of AKA under the division of IHCS or lay volunteers of Aberdeen Kai-fong Welfare Association volunteer group

Exclusion criteria

* Subjects refuse to answer this questionnaire
* Subjects who are unable to read and understand Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Staff of AKA under the division of IHCS or lay volunteers of Aberdeen Kai-fong Welfare Association volunteer group
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Perceived usefulness on institutional risk management | Baseline
  Measured by 15 outcome-based questions. Score of each question ranges from 1 to 6. The highest scores the better the outcomes.
Change from baseline competence in delivering health-related information and service to service users | Baseline, immediate after workshop
  Measured by 4 outcome-based questions. Score of each question ranges from 0 to 10. The highest scores the better the outcomes.

SECONDARY OUTCOMES:
Change in baseline competence in delivering health-related information at month1 | Baseline, month 1
  Measured by 4 outcome-based questions. Score of each question ranges from 0 to 10.
Change in baseline competence in delivering health-related information at month 3 | Baseline, month 3
  Measured by 4 outcome-based questions. Score of each question ranges from 0 to 10.
Change in baseline practice in delivering health-related information at month1 | Baseline, month 1
  Measured by a outcome-based question. Score of each question ranges from 0 to 10.
Change in baseline practice in delivering health-related information at month 3 | Baseline, month 3
  Measured by a outcome-based question. Score of each question ranges from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Abedreen Kai-fong Association, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Need to obtain consent from participants before agreeing to share individual participants data.
Supporting Information: Study Protocol
Time Frame: When study finished
Access Criteria: The minimal anonymized dataset will be available upon request to interested researchers. For interested researchers, please contact Dr Agnes Lai (Email: agneslai@hku.hk, School of Nursing, the University of Hong Kong), for further information.

REFERENCES:
- [Background] Rowe TA, Patel M, O'Conor R, McMackin S, Hoak V, Lindquist LA. COVID-19 exposures and infection control among home care agencies. Arch Gerontol Geriatr. 2020 Nov/Dec;91:104214. doi: 10.1016/j.archger.2020.104214. Epub 2020 Jul 30. PMID 32768800
- [Background] Pearce J, Mann MK, Jones C, van Buschbach S, Olff M, Bisson JI. The most effective way of delivering a train-the-trainers program: a systematic review. J Contin Educ Health Prof. 2012 Summer;32(3):215-226. doi: 10.1002/chp.21148. PMID 23173243
- [Background] Quandt SA, Grzywacz JG, Talton JW, Trejo G, Tapia J, D'Agostino RB Jr, Mirabelli MC, Arcury TA. Evaluating the effectiveness of a lay health promoter-led, community-based participatory pesticide safety intervention with farmworker families. Health Promot Pract. 2013 May;14(3):425-32. doi: 10.1177/1524839912459652. Epub 2012 Oct 17. PMID 23075501
- [Background] Ayala GX, Vaz L, Earp JA, Elder JP, Cherrington A. Outcome effectiveness of the lay health advisor model among Latinos in the United States: an examination by role. Health Educ Res. 2010 Oct;25(5):815-40. doi: 10.1093/her/cyq035. Epub 2010 Jul 5. PMID 20603384
- [Background] Shiber S, D'Lugoff M. A win-win model for an academic nursing center: community partnership faculty practice. Public Health Nurs. 2002 Mar-Apr;19(2):81-5. doi: 10.1046/j.1525-1446.2002.19202.x. PMID 11860592
- [Background] Josiah Willock R, Mayberry RM, Yan F, Daniels P. Peer training of community health workers to improve heart health among African American women. Health Promot Pract. 2015 Jan;16(1):63-71. doi: 10.1177/1524839914535775. Epub 2014 Jun 2. PMID 24891525
- [Background] Tobias CR, Downes A, Eddens S, Ruiz J. Building blocks for peer success: lessons learned from a train-the-trainer program. AIDS Patient Care STDS. 2012 Jan;26(1):53-9. doi: 10.1089/apc.2011.0224. Epub 2011 Nov 21. PMID 22103430
- [Background] Layne JE, Sampson SE, Mallio CJ, Hibberd PL, Griffith JL, Das SK, Flanagan WJ, Castaneda-Sceppa C. Successful dissemination of a community-based strength training program for older adults by peer and professional leaders: the people exercising program. J Am Geriatr Soc. 2008 Dec;56(12):2323-9. doi: 10.1111/j.1532-5415.2008.02010.x. PMID 19112654
- [Background] Milburn K. A critical review of peer education with young people with special reference to sexual health. Health Educ Res. 1995 Dec;10(4):407-20. doi: 10.1093/her/10.4.407. PMID 10159674
- See also: Life expectancy at birth, total (years)- Hong Kong SAR, China — https://data.worldbank.org/indicator/SP.DYN.LE00.IN?locations=HK]
- See also: Hospital discharges to home health rebounding — https://avalere.com/press-releases/hospital-discharges-to-home-health-rebound-while-snf-volumes-lag